CLINICAL TRIAL: NCT04247750
Title: Treatment of Beta-thalassemia Patients With Rapamycin (Sirolimus): From Pre-clinical Research to a Clinical Trial" - "Trattamento di Pazienti Con Beta-talassemia Con Rapamicina (Sirolimus): Dalla Ricerca Pre-clinica ad Uno Studio Clinico
Brief Title: Testing SIROLIMUS in Beta-thalassemia Transfusion Dependent Patients (THALA-RAP)
Acronym: THALA-RAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Rare Partners srl Impresa Sociale (Other); Meyer Children's Hospital IRCCS (Other); Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Maria Rita Gamberini, Medical Director, Azienda USL Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-001469-18 (EudraCT num)
Record Dates: First submitted 2020-01-08; First posted 2020-01-30 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Beta-Thalassemia
Keywords: rapamycin; erythroid differentiation; γ-globin; fetal haemoglobin
MeSH Terms: conditions — beta-Thalassemia | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Interventional, pilot, open-label phase II study with sirolimus in patients with transfusion-dependent beta-thalassemia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label trial (Experimental): Sirolimus 0.5 mg tablets
  Interventions: Drug: Sirolimus 0.5 mg

INTERVENTIONS:
Drug: Sirolimus 0.5 mg — Daily administration of 1 or more tablets

SUMMARY:
In β-thalassaemia and Sickle Cell Disease (SCD), a significant production of fetal haemoglobin (HbF) may reduce the severity of clinical course and reactivation of γ-globin gene expression in adulthood. HbF induction is one of the best strategies to ameliorate the characteristic symptoms of these diseases. Hydroxyurea (HU) is the only medication, approved by the US Food and Drug Administration, inducing HbF. However, treatments with HU induce sufficient HbF levels in only half of the patients, and side effects including leukopenia and neutropenia are frequently reported. Therefore, novel therapeutic inducers must be identified to develop a personalized treatment in β-thalassaemia and sickle cell anaemia. The availability of new treatments depends on drugs already approved for other indications, and on pharmacokinetics and pharmacovigilance already assessed. Rapamycin (as Sirolimus) is an immunosuppressant agent, approved by the FDA for acute rejection prevention in renal transplant recipients. The ability of this drug to induce γ-globin gene expression in erythroleukemia cell line and erythroid precursors cells (ErPCs) in ß-thalassaemia patients is already known. A clinical investigation on the effects of sirolimus in ß-Thalassaemia aims to evaluate several parameters related to red blood cell status and HbF levels and is a first step for the full clinical development in this new indication.

DETAILED DESCRIPTION:
The general aim of this protocol is to demonstrate the applicability of a personalised and precision medicine approach in beta-thalassaemia; the clinical trial setting repurposes a drug, namely sirolimus. The presence of high Fetal Hemoglobin (HbF) levels is considered a condition predictive of a favourable outcome in thalassaemia. Its increase induced by pharmacological agents is considered a potential way to improve the clinical status of the patients. In terms of efficacy analysis, the investigators will focus their attention on HbF levels.

Primary objective:

• The suitability evaluation of sirolimus for the treatment of beta-thalassemia patients within the frame of a comprehensive project aimed at the reduction of their transfusions need, with consequent amelioration of their quality of life. The purpose can be achieved through increasing of HbF levels pharmacologically mediated, with verification of a prerequisite, namely the correlation between the induction of HbF in vitro and in vivo in single patients.

Secondary objectives:

* To assess the safety of sirolimus and correlation between administered dose and blood levels in beta-thalassemia patients
* To assess the influence of sirolimus on transfusion regimen
* To assess the effect of sirolimus on the hematopoietic and immune system of thalassemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age;
* Patients able to understand the informed consent and to sign it before any study procedure;
* Patients with β0/β0 and β+/β0 thalassaemia genotype;
* Documented diagnosis of major or intermediate thalassemia transfusion-dependent (number of transfusions not less than 8 over the past 12 months before selection);
* On regular transfusion since at least 6 years;
* Splenectomy performed at least 60 days before selection or spleen largest dimensions < 20 cm as detected by abdominal echography;
* Female participants who are surgically sterilised/hysterectomised or post-menopausal for longer than 2 years or female participants of childbearing potential using and/or willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or using any other method considered sufficiently reliable by the investigator in individual cases. Patients must be counselled concerning measures to be used to prevent pregnancy and potential toxicities prior to the first dose of sirolimus;
* Patient willing to follow all the study requirements and perform all the study visits and to cooperate with the investigator;
* Patient followed by the same clinical site since at least 6 months.

Note that patients will be treated with oral sirolimus only in the case their Erythroid Precursor Cells (ErPCs) are responsive to the in vitro treatment with sirolimus according to laboratory-specific definition (≥ 20% increase of HbF in comparison with samples not treated with sirolimus);

Exclusion Criteria:

* Patient treated with hydroxyurea at selection visit or in the last 6 months;
* Ongoing treatment with drugs possibly affecting sirolimus actions;
* Documented aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x Upper Limit of Normal (ULN) at selection;
* Documented Platelet count <150.000/microliter and >1.000.000/microliter at selection;
* Heart failure as classified by the New York Heart Association (NYHA) classification 3 or higher;
* Uncontrolled hypertension defined as systolic blood pressure (BP) ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg;
* Significant arrhythmia requiring treatment,
* Corrected QT interval> 450 msec on selection ECG;
* Ejection fraction <50% by echocardiogram, multiple gated acquisition scan or cardiac magnetic resonance;
* Myocardial infarction within 6 months prior to selection;
* Positivity for human immunodeficiency virus (HIV) antibody, active hepatitis B (HBV) or hepatitis C (HCV) as demonstrated by the presence of hepatitis B surface antigen (HBsAg) and a positive HCV-RNA test, HBcAb and HBV-DNA positivity
* White blood cell [WBC] count <3000 cells per μL and/or Granulocytes <1500/mm3;
* Total cholesterol > 240 mg/dl;
* Triglycerides > 200 mg/dl;
* Proteinuria with urinary protein >1g/24 hrs;
* Current participation in another trial with an investigational drug or experimental device, or inclusion in another trial with an investigational drug or experimental device within the preceding month;
* Major surgery (including splenectomy) within 60 days before selection (patients must have fully recovered from any previous surgery);
* Iron chelation therapy changed in the last 3 months prior to selection (note that Deferiprone is not accepted as a chelation therapy drug in this study while Desferrioxamine and Deferasirox are tolerated at stable dose);
* Current treatment with macrolide antibiotics (clarithromycin);
* Pregnant or lactating women;
* History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the experimental drug;
* Treatment with live vaccines within 90 days preceding the selection;
* Subject with history or current malignancies (solid tumours and haematological malignancies) or presence of masses/tumour detected by ultrasound at selection;
* Subject with any significant medical condition and/or laboratory abnormality considered by the investigator as not adequately controlled at the time of selection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of fetal hemoglobin level | 360 days
  Fetal hemoglobin level in peripheral blood at day 360 compared to day 0, assessed through high pressure liquid chromatography (HPLC)

SECONDARY OUTCOMES:
Change from baseline of fetal hemoglobin level | 90-180 days
  Fetal hemoglobin level in peripheral blood at days 90 and 180 compared to day 0, assessed through HPLC
Change from baseline of γ-globin expression | 90-180-360 days
  Level of induction of the γ-globin expression at day 90, 180 and 360 compared to day 0
Change from baseline of biomarkers for erythropoiesis | 180-360 days
  - Evaluation of the Reticulocytes number at day 180 and 360 compared to baseline.
Change from baseline of biomarkers for erythropoiesis | 180-360 days
  - Evaluation of the Nucleated red blood cells number at day 180 and 360 compared to baseline.
Change from baseline of biomarkers for erythropoiesis | 180-360 days
  - Evaluation of the erythropoietin level at day 180 and 360 compared to baseline.
Change from baseline of biomarkers for erythropoiesis | 180-360 days
  - Evaluation of the serum transferrin receptor level at day 180 and 360 compared to baseline.
Change from baseline of biomarkers for haemolysis | 180-360 days
  - - Evaluation of the biomarkers for haemolysis level at day 180 and 360 compared to baseline. Biomarkers will include: serum bilirubin level
Change from baseline of biomarkers for haemolysis | 180-360 days
  - - Evaluation of the biomarkers for haemolysis level at day 180 and 360 compared to baseline. Biomarkers will include: serum lactate dehydrogenase (LDH) level
Change from baseline of tranfusion needs | 360 days
  Measurement of the total blood quantity (in mL) transfused (day -360 to -180, day -180 to 0, day 0 to 180, day 180 to 360)
Change from baseline of tranfusion needs | 360 days
  Recording of the number of transfusions done in a semester (day -360 to -180, day -180 to 0, day 0 to 180, day 180 to 360)
Change from baseline of Iron status | 180-360 days
  • Evaluation of the intake of iron chelators at days 180 and 360 compared to baseline
Change from baseline of Iron status | 90-180-360 days
  • Evaluation of serum ferritin level at day 90, 180 and 360 in comparison with day 0
Change from baseline of Immune function | 90-360 days
  • Peripheral blood immunophenotype-Lymphocyte subsets at day 90 and 360 compared to day 0
Change from baseline of Immune function | 90-360 days
  • Quantitative analysis of ImmunoglobulinG/ImmunoglobulinA/ImunoglobulinM at day 90 and 360 compared to day 0
Change from baseline of Quality of Life | 360 days
  Evaluation of the patient quality of life at 6 and 12 months compared to baseline through Transfusion-dependent Quality of Life questionnaire (TranQol), measuring specifically the quality of life in patients with thalassemia. The TranQol is a disease-specific Quality of Life measure that has been shown to be valid and reliable (Klaassen et al, British Journal of Haematology, 2014, 164, 431-437). On a total scale of 0-100, higher values always represent a better outcome. The questions are grouped into four domains: physical health, emotional health, family functioning, and school and career functioning. The adult self-report questionnaires include a fifth category on sexual activity which is only one item. Subscales are summed

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - University of Ferrara Department of Life Sciences and Biotechnology, Ferrara, FE
  - Day Hospital Thalassaemia and Haemoglobinopathies (DHTE) - Azienda Ospedaliero-Universitaria S.Anna of Ferrara, Ferrara, FE
  - Thalassemia and Hemoglobinopathies Center Azienda Ospedaliero Universitaria Meyer, Florence, Fi
  - Pediatric oncohematology Azienda Ospedaliero Universitaria Pisana Ospedale Santa Chiara, Pisa, Pi

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study the study protocol and the clinical trial report will be available to other researchers. Publication of the data is planned
Supporting Information: Study Protocol
Time Frame: After completion of the Clinical Study Report preparation
Access Criteria: Free availability of the publication. Free availability of the study protocol upon request